CLINICAL TRIAL: NCT04347668
Title: Can Virtual Reality Reduce Depression and Agitation in Older Adults With Moderate to Severe Dementia? A Randomized Controlled Trial.
Brief Title: Can Virtual Reality Reduce Depression and Agitation in Older Adults With Moderate to Severe Dementia?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO 0032743
Record Dates: First submitted 2019-09-19; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-08

CONDITIONS: Moderate Dementia; Severe Dementia
Keywords: Depression; Agitation
MeSH Terms: conditions — Dementia; Depression; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial, VR will be compared to usual care for residents with moderate to severe dementia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): All residents are seen by a RN, with care by Registered Practical Nurse (RPN) and Personal Support Worker (PSW) staff 24/7. Residents supported by behavior support Ontario staff; include Behavior responsive team. Residents prior to admission have been assessed by the Geriatric program. Residents may receive psychotropic or cognitive enhancement medications. The residents are seen routinely seen once a week by the physician. Their Dementia is monitored weekly but the physician as well as daily by the registered staff. Quarterly or more frequently cognitive assessments are completed and referrals made to appropriate specialists. A day would include meals, engagement in scheduled and non-scheduled programs such as exercise, and activities, groups. Residents are supported in their activities of daily living, and social engagement. Specific interventions based on resident needs are supported in a Dementia capable environment.
  Interventions: Other: Usual Care
- Virtual Reality (Experimental): Virtual Reality (VR) is a scenario that simulates experiences. The immersive environment is similar to the real world, creating an experience. A person using virtual reality equipment is able to "look around" the artificial world, move around in it, and interact with virtual features or items. VR requires the user to use a multi-projected in their own room using BroomX to generate realistic images, sounds that simulate a user's physical presence in a virtual or imaginary environment. A library has been developed, set to music, as well, we will use library items already part of the BroomX. We will attempt to use BroomX in their own room or in a suitable room within the LTC home. The participants still get the immersive experience, and the projection device has automatic controls that conform the visuals to a 360 experience no matter what size the room is, or what chairs, window blinds, are in the room.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — VR requires the user to use a multi-projected in their own room using BroomX to generate realistic images, sounds and other sensations that simulate a user's physical presence in a virtual or imaginary environment
  Other Names: BroomX
  Arms: Virtual Reality
Other: Usual Care — meals, engagement in scheduled and non-scheduled programs such as exercise, and activities, groups. Residents are supported in their activities of daily living, and social engagement. Specific interventions based on resident needs are supported in a Dementia capable environment.
  Arms: Usual Care

SUMMARY:
Dementia is a term used to describe a collection of symptoms including memory loss, problems with reasoning and communication, and a reduction in a person's ability to carry out daily activities. The most common types of dementia are: Alzheimer's disease, vascular dementia, mixed dementia and dementia with Lewy bodies. Clinicians and families are looking for ways to deal with this challenging group of diseases to improve quality of life, reduce depression and agitation for individuals in long term care (LTC).

There are a variety of non-pharmacologic interventions for dementia often used in addressing physiological and behavioral challenges, new to this category of treatment is virtual reality (VR).

Virtual reality has been studied in mild cognitive impairment. Colleagues completed a systematic review of non-pharmacological intervention to treat older people with dementia and found music to be the only intervention effective, VR was not included as no studies were found.

The Registered Nurses Association of Ontario report non-pharmacological approaches are an important alternative to the use of antipsychotic medications. They recommend health-care providers should consider non-pharmacological interventions wherever possible as a first-line approach to the management of BPSD.

Virtual reality as proposed in this research will include music, library items will be selected that are person specific, and will provide sensory stimulation. To date there is no published research on the use the VR in moderate to severe dementia in LTC, looking at depression.

DETAILED DESCRIPTION:
Dementia is a term used to describe a collection of symptoms including memory loss, problems with reasoning and communication, and a reduction in a person's ability to carry out daily activities such as washing, dressing and cooking. The most common types of dementia are: Alzheimer's disease, vascular dementia, mixed dementia and dementia with Lewy bodies. Dementia is a progressive condition, which means that the symptoms will gradually get worse. Clinicians and families are looking for ways to deal with this challenging group of diseases to improve quality of life, reduce depression and agitation that often accompany dementia as it progresses and individuals are placed in long term care (LTC).

There are a variety of non-pharmacologic interventions for dementia ranging from traditional interventions such as behavioral therapy to newer interventions such as multisensory therapy. Often used in addressing physiological and behavioral challenges, some interventions have been shown to aid cognitive ability as well. "Cognitive stimulation," is a catchall term referring to non-pharmacologic interventions with a cognitive focus, new to this category of treatment is virtual reality (VR).

Virtual reality has been studied in mild cognitive impairment. A systematic review of studies evaluating computerized cognitive training and virtual reality cognitive training interventions for individuals at high risk of cognitive decline called mild cognitive decline documented consistent improvement in the domains of attention, executive function, visual and verbal memory, and also on the psychological symptoms of depression, anxiety, and apathy in participants. Colleagues completed a systematic review of non-pharmacological intervention to treat older people with dementia and found music to be the only intervention effective, VR was not included as no studies were found.

The Registered Nurses Association of Ontario completed a best practice guideline on Dementia based on current evidence in 2016. They report non-pharmacological approaches are an important alternative to the use of antipsychotic medications, which historically have been overused as a first-line strategy for managing behavioural and psychological systems of dementia (BPSD). They recommend health-care providers should consider non-pharmacological interventions wherever possible as a first-line approach to the management of BPSD.

The most well-studied and effective non-pharmacological approaches include listening to music/music therapy, effective communication and person-centred approaches and other sensory stimulation. Virtual reality as proposed in this research will include music, specific library items will be selected that are person specific, and will provide sensory stimulation in keep with the RNAO guidelines. To date there is no published research on the use the VR in moderate to severe dementia in LTC looking at depression as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Resident of Henley Place, Henley House, and Burton Manor
2. Cognitive Performance Scale score between 3 to 5.

Exclusion Criteria:

1. Without a medical diagnosis of dementia,
2. Diagnosis of epilepsy,
3. Those who are blind,
4. Residents at end of life,
5. Unable to communicate in English,
6. Residents whose substitute decision-maker is from the Public Trustee and Guardian office of Ontario.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-27 (Estimated)

PRIMARY OUTCOMES:
Cornell Scale for Depression | This will be completed weekly to compare this to the change from baseline over a 2 week period.
  The Cornell Scale for Depression is a 19 item scale that measures depression where a score of 12 or above indicates probable depression.

SECONDARY OUTCOMES:
The Cohen Mansfield Agitation Inventory | This will be completed weekly to compare this to the change from baseline over a 2 week period.
  The Cohen-Mansfield Agitation Inventory (CMAI; (Cohen-Mansfield and Kerin, 1986)) is a 29-item tool (Cohen-Mansfield et al., 1989) developed to assess agitated behaviours of people residing within nursing homes.
Percentage Sleep | This will be completed weekly to compare this to the change from baseline over a 2 week period.
  This is currently recorded in the participants electronic chart by the night staff.
Psychotropic medication | This will be completed weekly to compare this to the change from baseline over a 2 week period.
  From the chart we will record the use of psychotropic medications, both regular dose and prn's
Weight | Weight will be recorded before and after the intervention to compare the change from baseline over a 2 month period.
  From the chart we will record the weights of the participants
1 to 1 staff | We will record from administrative data the hours of 1 to 1 staff per participant, for 1 month, before and after the intervention. This will be completed monthly to compare this to the change from baseline over a 2 month period.
  We will record the number of hours of 1 to 1 staff usage to manage behaviours.
Transfers to the emergency department (ED) | We will record from the chart the transfer to the emergency department per participant, for 1 month, before and after the intervention. This will be completed monthly to compare this to the change from baseline over a two month period.
  From the chart we will record and transfers to the ED for catastrophic behaviours.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Burton Manor, Brampton, Ontario
  - Henley Place, London, Ontario
  - Henley House, Saint Catherines, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen-Mansfield J. Agitated behaviors in the elderly. II. Preliminary results in the cognitively deteriorated. J Am Geriatr Soc. 1986 Oct;34(10):722-7. doi: 10.1111/j.1532-5415.1986.tb04303.x. PMID 3760436
- [Result] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862